CLINICAL TRIAL: NCT06126900
Title: Smartphone App-assisted Short-term Antibiotic Therapy - a Cluster-randomized Study in Primary Care
Brief Title: Smartphone App-assisted Short-term Antibiotic Therapy
Acronym: SMAPP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 2023-01753
Record Dates: First submitted 2023-10-17; First posted 2023-11-13 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2025-01

CONDITIONS: Infection, Bacterial
Keywords: Medication Adherence; Short-term therapy; Anti-Bacterial Agents; Mobile Health
MeSH Terms: conditions — Bacterial Infections; Medication Adherence

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Reminder + text messaging
  Interventions: Other: Smartphone medication intake reminder + educational and motivational text messaging
- Control Group (No Intervention): No reminder + no text messaging

INTERVENTIONS:
Other: Smartphone medication intake reminder + educational and motivational text messaging — The intervention includes the use of a smartphone-based medication intake reminder, along with two educational and motivational text messages during the therapy period.
  Arms: Intervention Group

SUMMARY:
Outpatients with short-term antibiotic treatment should start and finish the treatment according to medical advise that is, the intake pattern (named adherence) should be regular. The research question is: Can a smartphone-based program including intake reminder and two text messages improve adherence to a short-term antibiotic treatment in ambulatory setting?

Participants will be asked to record every antibiotic intake in an app on their smartphone over the prescribed therapy duration and to note their symptoms once daily. One group will obtain reminder + text messages, and the control group will have no reminder + no text messages.

DETAILED DESCRIPTION:
This study is planned as a monocentric, cluster-randomized, double-blind, two-arm study in a primary care setting with outpatients newly prescribed co-amoxicillin for a short-term therapy. Participating community pharmacies will recruit patients entering with a prescription for co-amoxicillin and offer the service. Randomisation will take place on the pharmacy level via computer generated list of numbers (1: with intervention; 2: with no intervention). Pharmacists and participants will not know that the intervention is not the app itself, but rather the combination of a reminder and text messages (= double-blind). The intervention will consist of the use of a smartphone reminder (e.g. alarm clock or a reminder app; a list with suitable examples will be given and patients will choose one of them) and two personalized motivational and educational text messages that will be sent by the pharmacy during the treatment duration. The control group will have no reminder and no text messages. All participants will use a simplified version of the freely available medication management app TOM to record their medication intake (= adherence measurement method). Participants in both groups will obtain a consultation driven by their adherence report with the study team at the end of the treatment to discuss their individual adherence data, their symptom course and well-being. After that, patients will receive a link to an online survey where they will evaluate their satisfaction with the service and the smartphone application. Participating pharmacists will be interviewed by the study team regarding their experience and satisfaction after the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* is min. 18 years old;
* is newly prescribed a co-amoxicillin treatment of 3-14 days;
* has symptoms that correspond to bacterial infection;
* accepts to use of one of the medication adherence application with reminder function from the provided list;
* accepts to use of the electronic monitoring application TOM™ during the study period;
* is capable of using the TOM™ application;
* signs the informed consent form;
* understands and speaks (Swiss) German.

Exclusion Criteria:

* in the opinion of the pharmacists, unlikely to comply with the study schedule or are unsuitable for any other reason.
* does not manage medication himself/herself
* already using a medication intake reminder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2024-01-15 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Adherence rates (in percent) | Up to 14 days (maximum therapy duration)
  Patients confirm every medication intakes in the app. The app will deliver time stamps. Based on these, taking, dosing and timing adherence will be calculated in percent.

SECONDARY OUTCOMES:
Persistence rate (in percent) | Up to 14 days (maximum therapy duration)
  Patients confirm every medication intakes in the app. The app will deliver time stamps. Based on these, persistence rate to the therapy will be calculated: [days with at least one dose / prescribed treatment days] × 100
Time to symptom control | Up to 14 days (maximum therapy duration)
  Patients will note in a diary their symptoms once daily. Time to symptom control will be calculated as number of days up to freedom of symptoms.
Pharmacists' satisfaction with the service including the app | 2 weeks after study completion
  Satisfaction will be assessed through semi-structured interviews and analyzed inductively.
Patients' satisfaction with the service including the app | 7 days after therapy completion
  Satisfaction will be assessed quantitatively in an online-survey on a 5-point Likert-scale. High values will indicate a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle Arnet, Dr. PD, Principal Investigator — University of Basel, Pharmaceutical Care Research Group
Locations (2):
- Switzerland (2):
  - TopPharm Hirschen Apotheke, Magden, Canton of Aargau
  - Greifen Apotheke, Basel, Canton of Basel-City